CLINICAL TRIAL: NCT02224287
Title: Assessment of Fluoroscopy Times With Surgeon Versus Technologist Control: A Prospective Randomized Trial
Brief Title: Assessment of Fluoroscopy Times With Surgeon Versus Technologist Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Caleb Nelson, Caleb Nelson MD, MPH, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00003145
Record Dates: First submitted 2014-08-20; First posted 2014-08-25 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2017-04

CONDITIONS: Urolithiasis; Kidney Stones
Keywords: Urolithiasis; Kidney Stones; Ureteroscopy; Fluoroscopy
MeSH Terms: conditions — Urolithiasis; Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fluoroscopy (Other): Technologist control of fluoroscopy Surgeon control of fluoroscopy
  Interventions: Procedure: Technologist control of fluoroscopy; Procedure: Surgeon control of fluoroscopy

INTERVENTIONS:
Procedure: Technologist control of fluoroscopy — Technologist control of fluoroscopy
Procedure: Surgeon control of fluoroscopy — Surgeon control of fluoroscopy

SUMMARY:
This is a prospective randomized trial to study the effect of assigning the control of the fluoroscopic x-ray activation to the surgeon as compared to the radiation technologist. Radiation exposure will be assessed from the collected data, fluoroscopy time, and dose parameters (cumulative absorbed dose and dose area product). From exposure data, entrance skin dose (ESD) and midline absorbed dose (MLD) will be calculated. The primary outcome in this study will be total fluoroscopy time for the procedure. A secondary outcome will be the ESD. The investigators will further analyze the contribution of clinical predictors (e.g. stone size/location) and procedural predictors on fluoroscopy times and ESD.

It is hypothesized that a 30% reduction in fluoroscopy time will occur when the operating surgeon is controlling the activation of the x-ray beam.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ureteroscopy for urolithiasis
* 5 years to 25 years old

Exclusion Criteria:

* Pregnant
* Less than 5 years old or older than 25 years old

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2013-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome in this study will be total fluoroscopy time for the procedure. | 1-5 hours
  The average duration of a ureteroscopy is 1-5 hours. At the completion of the surgery, the individual outcomes will be assessed.

SECONDARY OUTCOMES:
A secondary outcome will be the entrance skin dose (mGy). We will further analyze the contribution of clinical predictors (e.g. stone size/location) and procedural predictors on fluoroscopy times and entrance skin dose. | 1-5 hours
  The average duration of a ureteroscopy is 1-5 hours. At the completion of the surgery, the individual outcomes will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Caleb Nelson, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kokorowski PJ, Chow JS, Cilento BG Jr, Kim DS, Kurtz MP, Logvinenko T, MacDougall RD, Nelson CP. The effect of surgeon versus technologist control of fluoroscopy on radiation exposure during pediatric ureteroscopy: A randomized trial. J Pediatr Urol. 2018 Aug;14(4):334.e1-334.e8. doi: 10.1016/j.jpurol.2018.04.035. Epub 2018 Jun 27. PMID 30257794